CLINICAL TRIAL: NCT02307968
Title: Comparison of Patient's Preference, Pain Perception, and Usability Between Inner and Outer Upper Thigh for Insulin Therapy
Brief Title: Comparative Study of Insulin Therapy Between Inner and Outer Upper Thigh
Acronym: CUSTIOT
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhou Weibin, MD, First Affiliated Hospital of Zhejiang University
Other Study IDs: ChiCTR-OPN-14005516
Record Dates: First submitted 2014-11-25; First posted 2014-12-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- inner thigh insulin injection: inject insulin at inner thigh site is the intervention arm. So we inject insulin at this site to see if this site is suitable for insulin injection.
  Interventions: Other: insulin injection site
- outer thigh insulin injection: outer thigh site for insulin therapy is the usual site

INTERVENTIONS:
Other: insulin injection site — insulin injected site between inner thigh and out thigh
  Groups: inner thigh insulin injection

SUMMARY:
To observe the patient's preference, pain perception, and usability between inner and outer upper thigh for insulin therapy. To add another injection site for insulin therapy.

DETAILED DESCRIPTION:
The most common injection site is the abdomen (or stomach). The back of the upper arms, the upper buttocks or hips, and the outer side of the thighs are also used. These sites are the best to inject into for two reasons: They have a layer of fat just below the skin to absorb the insulin, but not many nerves - which means that injecting there will be more comfortable than injecting in other parts of your body. But while the needle for insulin therapy is becoming shorter, it is possible to inject insulin at the inner thigh site.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients more than 18 years age old with diabetes that need insulin therapy

Exclusion Criteria:

* Those diabetes with psychologic diseases and those patients won't be injected at thigh

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetes population
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
pain | immediately after injection, 1-5minutes
  the pain degree the patient feel while insulin injected using Visual Analog scale
bleeding | immediately after injection, 1-5minutes
  if bleeding occurs after insulin injected just by using Yes or No
leaking | immediately after injection, 1-5minutes
  if there is leaking after insulin injected just by using Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Jingyun Yuan, BS, Principal Investigator — Department of Endocrinology, the First Affiliated Hospital to Zhejiang University School of Medicine
Locations (1):
- Department of Endocrinology, the First Affiliated Hospital to Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Yuan J, Chen Y, Xuan Y, Cao L, Zhu J, Wang F, Zhou X, Ye Q, Liao L, Zheng Y, Zhou Q, Chen X, Chen M, Zhou W. Can the upper inner side of the thigh become a new option for insulin injection? Curr Med Res Opin. 2016 Jul;32(7):1319-24. doi: 10.1185/03007995.2016.1174107. Epub 2016 May 17. PMID 27090917